CLINICAL TRIAL: NCT01841307
Title: Development and Validation of Test for Gastro-esophageal Reflux and Aspiration
Brief Title: Cromolyn Detection of Silent Aspiration
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Difficulty recruiting; Funding ended; interim analysis provided sufficient data for interpretation.
Sponsor: University of California, San Francisco (Other)
Collaborators: Aradign Corportation (Unknown); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-11080
Record Dates: First submitted 2013-04-23; First posted 2013-04-26 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Gastroesophageal Reflux; Respiratory Aspiration; Idiopathic Pulmonary Fibrosis; Lung Transplantation
MeSH Terms: conditions — Gastroesophageal Reflux; Respiratory Aspiration; Idiopathic Pulmonary Fibrosis | interventions — Cromolyn Sodium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gastrocrom (Experimental): 4 ingestions (at 2h intervals) of a 200 mL of a 1mg/mL solution of cromolyn sodium (inpatient) OR 2 ingestions (at 4h intervals) of a 200 mL of a 1mg/mL solution of cromolyn sodium (outpatient)
  Interventions: Drug: Cromolyn Sodium

INTERVENTIONS:
Drug: Cromolyn Sodium
  Other Names: Gastrocrom

SUMMARY:
The overall purpose of this project is to develop and validate a simple, non-invasive method to detect aspiration of gastro-intestinal fluid into the respiratory tract. In the inpatient setting, the investigators will compare the quantity of cromolyn detected in urine collected overnight after 4 ingestions (at 2h intervals) of a 200 mL of a 1mg/mL solution of cromolyn sodium, by 5 healthy control subjects and 5 patients (3-6 with pulmonary fibrosis; and 3-6 either awaiting or recently undergone lung transplantation) with clinical and laboratory evidence of GER (gastroesophageal reflux) with microaspiration. In the outpatient setting, the investigators will compare the quantity of cromolyn detected in urine collected overnight after 1 ingestions (at 4h intervals) of a 200 mL of a 1mg/mL solution of cromolyn sodium, by 10 patients (3-6 with pulmonary fibrosis; and 3-6 either awaiting or recently undergone lung transplantation) with clinical and laboratory evidence of GER (gastroesophageal reflux) with microaspiration.

ELIGIBILITY:
Inclusion Criteria:

Healthy participants

* Adult non-smokers
* Females only - negative urine pregnancy test

Lung transplant patients

* Adult patients awaiting (or recently undergone) - lung transplant
* Evidence of gastro-esophageal reflux with probable recurrent aspiration
* Females only - negative urine pregnancy test

Idiopathic pulmonary fibrosis patients

* Adult patients currently enrolled in on-going University of California, San Francisco study of prevalence of recurrent GER with aspiration in idiopathic pulmonary fibrosis
* Evidence of gastro-esophageal reflux with probable recurrent aspiration
* Females only - negative urine pregnancy test

Exclusion criteria:

Healthy participants

* History of dysphagia
* GER
* Recurrent cough
* Asthma
* Pneumonia after childhood
* Sleep impairment
* Use of drugs or alcohol impairing consciousness
* Impaired gag reflex on physical examination
* Any other significant medical illness (e.g., morbid obesity, diabetes, neurologic disease, etc.) that in the opinion of the investigator could affect the clinical features measured, responses to the therapies to be given in this study, or risks of participating in the study
* Greater than 5 pack years lifetime smoking history
* History of intolerance or allergy to cromolyn sodium

Lung transplant patients

* History of intolerance or allergy to cromolyn sodium
* History of Nissen fundoplication

IPF patients

* History of intolerance or allergy to cromolyn sodium
* History of Nissen fundoplication

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Total cromolyn in urine collected overnight | Collected overnight (6 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Homer Boushey, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Airway Clinical Research Center, San Francisco, California, United States